CLINICAL TRIAL: NCT05213624
Title: A Multicenter, Randomized, Double-blind, Parallel Group, Placebo-controlled Study to Assess the Efficacy, Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Profile of BI 764198 Administered Orally Once Daily for 12 Weeks in Patients With Focal Segmental Glomerulosclerosis
Brief Title: A Study to Test BI 764198 in People With a Type of Kidney Disease Called Focal Segmental Glomerulosclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1434-0004; 2020-000384-23 (EudraCT Number); U1111-1292-1333 (Registry Identifier: UTN, WHO registry)
Record Dates: First submitted 2022-01-27; First posted 2022-01-28 (Actual); Results first posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Kidney Disease, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BI 764198 20 mg (Experimental): Patients with primary focal segmental glomerulosclerosis (FSGS) or patients with monogenic FSGS as a result of TRPC6 mutations took daily one single capsule of 20 milligrams (mg) of BI 764198 orally for 12 weeks.
  Interventions: Drug: BI 764198
- BI 764198 40 mg (Experimental): Patients with primary focal segmental glomerulosclerosis (FSGS) or patients with monogenic FSGS as a result of TRPC6 mutations took daily one single capsule of 40 milligrams (mg) of BI 764198 orally for 12 weeks.
  Interventions: Drug: BI 764198
- BI 764198 80 mg (Experimental): Patients with primary focal segmental glomerulosclerosis (FSGS) or patients with monogenic FSGS as a result of TRPC6 mutations took daily one single capsule of 80 milligrams (mg) of BI 764198 orally for 12 weeks.
  Interventions: Drug: BI 764198
- Placebo (Placebo Comparator): Patients with primary focal segmental glomerulosclerosis (FSGS) or patients with monogenic FSGS as a result of TRPC6 mutations took daily one single capsule of placebo-matching BI 764198 orally for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 764198 — One single capsule of 20 milligrams (mg), 40 mg, or 80 mg of BI 764198 orally, once a day.
  Arms: BI 764198 20 mg; BI 764198 40 mg; BI 764198 80 mg
Drug: Placebo — One single capsule of placebo matching BI 764198 orally, once a day.
  Arms: Placebo

SUMMARY:
This study is open to adults with a type of kidney disease called focal segmental glomerulosclerosis (FSGS). The purpose of this study is to find out whether a medicine called BI 764198 improves the health of the kidneys in people with FSGS. Three different doses of BI 764198 are tested in this study.

Participants are put into 4 groups randomly, which means by chance. Three of the groups receive different doses of BI 764198 and one group receives placebo. Participants are in the study for about 4 months. For about 3 months, they take BI 764198 or placebo as capsules once a day.

Placebo capsules look like BI 764198 capsules but do not contain any medicine. Participants visit the study site about 10 times. You can participate in this study from your home. In this case a research nurse will visit you for the study visits.

Kidney health is assessed based on the analysis of urine samples, which participants collect at home. At the end of the study, the results are compared between the different groups. During the study, the doctors also regularly check the general health of the participants.

ELIGIBILITY:
Inclusion criteria:

* Male and female patients 18 years to 75 years (both inclusive) of age on the day of signing informed consent.
* Patients diagnosed with biopsy proven primary Focal Segmental Glomerulosclerosis (FSGS) or documented Transient Receptor Potential Cation subfamily C Member 6 (TRPC6) gene mutation causing FSGS prior to screening visit.
* Urine Protein-Creatinine Ratio (UPCR) ≥ 1000 mg/g based on first morning void urine sample during screening.
* Patients treated with corticosteroids must be on a stable dose for at least 4 weeks prior to screening visit with no plan to change the dose until end of trial treatment.
* Patients treated with Angiotensin Converting Enzyme (ACE) inhibitors, Angiotensin II Receptor Blockers (ARBs), finerenone, aldosterone inhibitors, or Sodium-Glucose Cotransporter-2 (SGLT2) inhibitors should be on a stable dose for at least 4 weeks prior to screening visit with no plan to change the dose until end of trial treatment.
* Body Mass Index (BMI) of ≤ 40 kg/m² at screening visit.
* Women of childbearing potential (WOCBP) must be willing and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the informed consent form (ICF) and in the study protocol.

Further inclusion criteria apply.

Exclusion criteria:

* Known monogenic (with the exception of TRPC6 gene mutations) or clinical or histologic evidence of secondary FSGS.
* Documented Alport syndrome, Nail Patella syndrome, diabetic nephropathy, Immunoglobulin A (IgA)-nephropathy, lupus nephritis, or monoclonal gammopathy (e.g., multiple myeloma).
* Concomitant use of calcineurin inhibitors.
* Concomitant treatment with cytotoxic agents (cyclophosphamide, chlorambucil), or CD20 monoclonal antibody, e.g., rituximab, within 5 half-lives before screening visit. Note: use of other immunosuppression therapies considered as standard of care may be allowed as long as the patient remains on stable dose throughout the study.
* Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m² at screening visit.
* Time between start of the Q-wave and end of the T-wave in an electrocardiogram interval corrected for heart rate (QTc) intervals (QT interval corrected for heart rate using the method of Fridericia - QTcF) greater than 450 ms in males or greater than 470 ms in females, or any other clinically relevant electrocardiogram (ECG) findings (at the investigator's discretion) at screening visit.
* Detection of graded cataract by Lens Opacities Classification System III (LOCS III) higher than NC1/NO1, C0, P0 in the slit lamp eye examination at screening visit. Planned cataract surgery during participation in the study. Patients with cataract who have undergone lens replacement are not excluded.
* Women who are pregnant, nursing, or who plan to become pregnant while in the study.

Further exclusion criteria apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-01-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (54):
- United States (20):
  - Nephrology Consultants, LLC, Huntsville, Alabama
  - University of California San Francisco, San Francisco, California
  - Valiance Clinical Research-South Gate-67878, South Gate, California
  - Valiance Clinical Research-Tarzana-68237, Tarzana, California
  - The Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Elixia Fort Lauderdale, LLC, Fort Lauderdale, Florida
  - South Florida Research Institute, Lauderdale Lakes, Florida
  - Total Research Group, LLC, Miami, Florida
  - Emory Children's Center, Atlanta, Georgia
  - NANI Research, LLC, Oak Brook, Illinois
  - University of Michigan Health System, Ann Arbor, Michigan
  - Jacobi Medical Center, The Bronx, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Texas Tech University Health Sciences Center-Amarillo-63885, Amarillo, Texas
  - Dallas Nephrology Associates Medical Clinic, DeSoto, Texas
  - Prolato Clinical Research Center-Houston-68087, Houston, Texas
- Australia (5):
  - Liverpool Hospital, Liverpool, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Griffith Health, Southport, Queensland
  - Sunshine Hospital, AT Albans, Victoria
- UZ Leuven, Leuven, Belgium
- China (8):
  - Fu Yang people's Hospital, Fuyang
  - Guangdong Provincial People's Hospital, Guangzhou
  - The First Afiliated Hospital, Sun Yet-sen University, Guangzhou
  - Zhejiang Province People's Hospital, Hangzhou
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The First People's Hospital of Nanning, Nanning
  - Tongren hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai Fifth People's Hospital affiliated to Fudan University, Shanghai
- France (3):
  - HOP Pellegrin, Bordeaux
  - HOP Bicêtre, Le Kremlin-Bicêtre
  - HOP Hôtel-Dieu, Nantes
- Germany (3):
  - Universitätsklinikum Köln (AöR), Cologne
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
- Italy (3):
  - A.O. Policlinico Giovanni XXIII di Bari, Bari
  - Policlinico S. Orsola-Malpighi, Bologna
  - Fondazione Salvatore Maugeri, Pavia
- New Zealand (2):
  - New Zealand Clinical Research (ChristChurch), Christchurch
  - Dunedin Hospital, Dunedin
- Spain (6):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital del Mar, Barcelona
  - Fundació Puigvert, Barcelona
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- United Kingdom (3):
  - St Luke's Hospital, Bradford
  - Addenbrooke's Hospital, Cambridge
  - Salford Royal, Salford

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Trachtman H, Kretzler M, Gesualdo L, Cross N, Workeneh B, Kaufeld J, Meijers B, Ye Z, Chen Q, Derebail VK, Ng MSY, Ji B, Lobmeyer MT, Retlich S, Licariao Rocha FT, Prasad S, Soleymanlou N. TRPC6 inhibition for the treatment of focal segmental glomerulosclerosis: a randomised, placebo-controlled, phase 2 trial of BI 764198. Lancet. 2026 Jan 27:S0140-6736(25)02255-X. doi: 10.1016/S0140-6736(25)02255-X. Online ahead of print. PMID 41616795
- [Derived] Wooden B, Beenken A, Martinelli E, Saida K, Knob AL, Ke J, Pisani I, Jin G, Lane B, Mitrotti A, Colby E, Lim TY, Guglielmi F, Osborne AJ, Ahram DF, Wang C, Armand F, Zanoni F, Bomback AS, Delsante M, Appel GB, Ferrari MRA, Martino J, Sahdeo S, Breckenridge D, Petrovski S, Paul DS, Hall G, Magistroni R, Murtas C, Feriozzi S, Rampino T, Esposito P, Helmuth ME, Sampson MG, Kretzler M, Kiryluk K, Shril S, Gesualdo L, Maggiore U, Fiaccadori E, Gbadegesin R, Santoriello D, D'Agati VD, Saleem MA, Gharavi AG, Hildebrandt F, Pollak MR, Goldstein DB, Sanna-Cherchi S. Natural History and Clinicopathological Associations of TRPC6-Associated Podocytopathy. J Am Soc Nephrol. 2025 Feb 1;36(2):274-289. doi: 10.1681/ASN.0000000501. Epub 2024 Oct 1. PMID 39352759
- [Derived] Salemkour Y, Yildiz D, Dionet L, 't Hart DC, Verheijden KAT, Saito R, Mahtal N, Delbet JD, Letavernier E, Rabant M, Karras A, van der Vlag J, Nijenhuis T, Tharaux PL, Lenoir O. Podocyte Injury in Diabetic Kidney Disease in Mouse Models Involves TRPC6-mediated Calpain Activation Impairing Autophagy. J Am Soc Nephrol. 2023 Nov 1;34(11):1823-1842. doi: 10.1681/ASN.0000000000000212. Epub 2023 Sep 6. PMID 37678257
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomized, double-blind, parallel group trial to assess the efficacy of 3 doses of BI 764198 (20 mg, 40 mg, and 80 mg) compared to placebo in patients with primary focal segmental glomerulosclerosis (FSGS), or patients with monogenic FSGS as a result of TRPC6 mutations.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | BI 764198 20 mg | BI 764198 40 mg | BI 764198 80 mg | Placebo
Started | 18 | 16 | 17 | 16
Treated | 18 | 15 | 15 | 14
Completed | 18 | 10 | 15 | 13
Not Completed | 0 | 6 | 2 | 3
Not completed — Adverse Event | 0 | 3 | 0 | 0
Not completed — Protocol deviation | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Not treated | 0 | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Treated set: all patients who received at least one dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 764198 20 mg | BI 764198 40 mg | BI 764198 80 mg | Placebo | Total
Number analyzed (Participants) | 18 | 15 | 15 | 14 | 62
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.2 (15.0) | 39.8 (13.8) | 39.8 (10.5) | 42.2 (11.1) | 40.7 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 2 | 7 | 25
  Male | 9 | 8 | 13 | 7 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 2 | 0 | 10
  Not Hispanic or Latino | 12 | 13 | 13 | 14 | 52
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 3 | 3 | 2 | 4 | 12
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 0 | 2
  Black or African American | 2 | 0 | 1 | 1 | 4
  White | 11 | 10 | 9 | 9 | 39
  More than one race | 1 | 2 | 1 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Urine Protein-Creatinine Ratio (UPCR) from 24-hour Urine [Mean (Standard Deviation); unit: Ratio] | 4.4865 (3.0188) | 4.0508 (3.0012) | 2.6767 (2.2209) | 4.5166 (2.9342) | 3.9709 (2.8565)

OUTCOME MEASURES:

1. Primary Outcome: Achievement of at Least 25% Reduction in 24-hour Urine Protein Creatinine Ratio (UPCR) Relative to Baseline at Week 12
Description: Predicted probability of patients as a percentage - predicted percentage of patients - achieving at least 25% reduction in 24-hour urine protein creatinine ratio (UPCR) relative to baseline at Week 12 (responders) is reported. Baseline was the average of two 24-hour urine samples collected before Visit 2 (Week 0). Patients who either missed their Week 12, 24-hour UPCR assessment or their Week 12, 24-hour UPCR assessment, occurred later than 5 days after the last dose (Residual Effect Period), were considered as non-responders.
  The predicted probability of response was calculated using a logistic regression utilizing corticosteroid use at randomization and baseline 24-hr UPCR as covariates and is presented as a percentage.
Time Frame: At baseline and Week 12.
Population: Full Analysis Set (FAS): all patients who were randomized and treated with evaluable measurements of 24-hr UPCR at baseline and at least one 24-hr UPCR measurement after the first dose. Patients who either missed their Week 12, 24-hour UPCR assessment or their Week 12, 24-hour UPCR assessment, occurred later than 5 days after the last dose (Residual Effect Period), were considered as non-responders and were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Predicted percentage of patients
Arm/Group | BI 764198 20 mg | BI 764198 40 mg | BI 764198 80 mg | Placebo
Number analyzed (Participants) | 18 | 14 | 14 | 14
Predicted percentage of patients | 48.9 [29.2 to 68.6] | 16.0 [-1.5 to 33.5] | 38.5 [12.2 to 64.8] | 11.4 [-2.3 to 25.2]
Statistical Analysis 1: Comparison: BI 764198 20 mg vs Placebo; Logistic regression utilizing corticosteroid use at randomization and baseline 24-hr UPCR as covariates; Test type: Other; Odds Ratio (OR) = 10.00, 95% CI 2-sided [1.59 to 118.14] — BI 764198 (comparator) vs. Placebo (reference)
Statistical Analysis 2: Comparison: BI 764198 40 mg vs Placebo; Logistic regression utilizing corticosteroid use at randomization and baseline 24-hr UPCR as covariates; Test type: Other; Odds Ratio (OR) = 1.53, 95% CI 2-sided [0.16 to 19.48] — BI 764198 (comparator) vs. Placebo (reference)
Statistical Analysis 3: Comparison: BI 764198 80 mg vs Placebo; Logistic regression utilizing corticosteroid use at randomization and baseline 24-hr UPCR as covariates; Test type: Other; Odds Ratio (OR) = 5.97, 95% CI 2-sided [0.86 to 73.57] — BI 764198 (comparator) vs. Placebo (reference)

2. Primary Outcome: Relative Change From Baseline at Week 12 of 24-hour Urine Protein Creatinine Ratio (UPCR)
Description: Relative change from baseline at Week 12 in 24-hour urine protein creatinine ratio (UPCR), is reported. Baseline was the average of two 24-hour urine samples collected before Visit 2 (Week 0).
  An analysis of covariance (ANCOVA) model was used to estimate the relative change in UPCR from baseline to Week 12 with corticosteroid use at randomization and baseline 24-hr UPCR as covariates.
Time Frame: At baseline and at Week 12.
Population: Full Analysis Set (FAS): all patients who were randomized and treated with evaluable measurements of 24-hr UPCR at baseline and at least one 24-hr UPCR measurement after the first dose. Patients who either missed their Week 12, 24-hour UPCR assessment or their Week 12, 24-hour UPCR assessment, occurred later than 5 days after the last dose (Residual Effect Period), were not included in this analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of change in 24-hour UPCR
Arm/Group | BI 764198 20 mg | BI 764198 40 mg | BI 764198 80 mg | Placebo
Number analyzed (Participants) | 16 | 10 | 13 | 11
Percentage of change in 24-hour UPCR | -38.44 [-50.41 to -23.60] | -2.39 [-24.50 to 26.19] | -21.52 [-39.18 to 1.27] | 2.28 [-20.20 to 31.09]
Statistical Analysis 1: Comparison: BI 764198 20 mg vs Placebo; An analysis of covariance (ANCOVA) model was used to estimate the change in UPCR from baseline to Week 12 with corticosteroid use at randomization and baseline 24-hr UPCR as covariates; Test type: Other; p = 0.0024, ANCOVA — Nominal and unadjusted; Relative difference = -39.82, 95% CI 2-sided [-56.17 to -17.36] — Comparison vs Placebo Calculated as (exp(difference of least square means) - 1) * 100
Statistical Analysis 2: Comparison: BI 764198 40 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.7906, ANCOVA — Nominal and unadjusted; Relative difference = -4.57, 95% CI 2-sided [-32.92 to 35.77] — Comparison vs Placebo Calculated as (exp(difference of least square means) - 1) * 100
Statistical Analysis 3: Comparison: BI 764198 80 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.1325, ANCOVA — Nominal and unadjusted; Relative difference = -23.27, 95% CI 2-sided [-45.83 to 8.70] — Comparison vs Placebo Calculated as (exp(difference of least square means) - 1) * 100

3. Secondary Outcome: Change in 24-hour Urine Protein Creatinine Ratio (UPCR) Relative to Visit 3 at Week 12
Description: Median change in 24-hour urine protein creatinine ratio (UPCR) relative to Visit 3 (Week 1) at Week 12, is calculated by subtracting the 24-hour UPCR, [Week 12] - [Week 1] values per patient, then by calculating the median of these changes, per treatment group.
Time Frame: At Week 1 and Week 12.
Population: Full Analysis Set (FAS): all patients who were randomized and treated with evaluable measurements of 24-hr UPCR at baseline and at least one 24-hr UPCR measurement after the first dose. Only patients with both a valid Visit 3 and Week 12, 24-hour UPCR value were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: grams/grams
Arm/Group | BI 764198 20 mg | BI 764198 40 mg | BI 764198 80 mg | Placebo
Number analyzed (Participants) | 15 | 10 | 12 | 10
grams/grams | -0.035 [-0.812 to 0.669] | 0.712 [-0.169 to 0.926] | -0.4435 [-0.837 to 0.1795] | 0.106 [-0.496 to 0.497]

4. Secondary Outcome: Change in 24-hour Urine Protein Creatinine Ratio (UPCR) Relative to Baseline at Week 13
Description: Median change in 24-hour urine protein creatinine ratio (UPCR) relative to baseline at Week 13, is calculated by subtracting the 24-hour UPCR, [Week 13] - [baseline] values per patient,then by calculating the median of these changes, per treatment group. Baseline was the average of two, 24-hour urine samples collected before Visit 2 (Week 0).
Time Frame: At baseline and at Week 13.
Population: Full Analysis Set (FAS): all patients who were randomized and treated with evaluable measurements of 24-hr UPCR at baseline and at least one 24-hr UPCR measurement after the first dose. Only patients with both a valid baseline and Week 13, 24-hour UPCR value were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: grams/grams
Arm/Group | BI 764198 20 mg | BI 764198 40 mg | BI 764198 80 mg | Placebo
Number analyzed (Participants) | 17 | 13 | 12 | 13
grams/grams | -0.4985 [-0.8080 to 0.5050] | -0.151 [-0.6945 to 0.7650] | -0.3033 [-0.5875 to 0.3830] | 0.0795 [-0.4410 to 1.4615]

5. Secondary Outcome: Change in 24-hour Urinary Protein Excretion Relative to Baseline at Week 12
Description: Median change in 24-hour urinary excretion rate relative to baseline at Week 12, is calculated by subtracting the urinary excretion rate, [Week 12] - [baseline], values per patient, then by calculating the median of these changes, per treatment group. Baseline was the average of two, 24-hour urine samples collected before Visit 2 (Week 0).
Time Frame: At baseline and at Week 12.
Population: Full Analysis Set (FAS): all patients who were randomized and treated with evaluable measurements of 24-hr UPCR at baseline and at least one 24-hr UPCR measurement after the first dose. Patients, who either missed their Week 12 urinary excretion rate measure or their Week 12 urinary excretion rate measure occurred later than 5 days after the last dose (Residual Effect Period), were not included in this analysis.
Measure: Median (Inter-Quartile Range); unit: grams/day
Arm/Group | BI 764198 20 mg | BI 764198 40 mg | BI 764198 80 mg | Placebo
Number analyzed (Participants) | 16 | 10 | 13 | 11
grams/day | -0.5036 [-1.6342 to -0.1112] | -0.4056 [-1.0535 to 0.6168] | -0.8967 [-1.0484 to -0.0975] | 0.0809 [-0.8115 to 1.7913]

6. Secondary Outcome: Pre-dose Plasma Concentration of BI 764198 at Steady-state (Cpre,ss ) at Week 4 and Week 12
Description: Pre-dose Plasma Concentration of BI 764198 at steady-state (Cpre,ss ) at Week 4 and Week 12 is reported.
Time Frame: At 671.917 hours and at 2015.917 hours after first drug administration.
Population: All patients who received at least one dose of trial medication and who provide at least one pre-dose concentration that was not excluded due to protocol violation relevant to the evaluation of pharmacokinetics (PK) or due to PK non-evaluability. Patients with no available pre-dose concentration were not included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/liter
Arm/Group | BI 764198 20 mg | BI 764198 40 mg | BI 764198 80 mg
Number analyzed (Participants) | 16 | 13 | 14
nanomole/liter
  Week 4: number analyzed (Participants) | 15 | 13 | 13
  Week 4 | 119 (47.2) | 266 (64.7) | 683 (66.5)
  Week 12: number analyzed (Participants) | 16 | 9 | 14
  Week 12 | 114 (85.9) | 328 (64.6) | 509 (45.7)

ADVERSE EVENTS:
Time Frame: All-cause mortality: From first drug-administration until individual end of trial. Up to approximately 16.4 weeks. Adverse event reporting: From first drug administration until stop of treatment + residual effect period (5 days). Up to 14 weeks.
Description: Treated set (TS): all patients who received at least one dose of trial medication.
Arm/Group | BI 764198 20 mg | BI 764198 40 mg | BI 764198 80 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/15 | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 3/18 | 0/15 | 1/15 | 1/14
Other Adverse Events (participants affected / at risk) | 14/18 | 10/15 | 10/15 | 10/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 764198 20 mg (N=18) | BI 764198 40 mg (N=15) | BI 764198 80 mg (N=15) | Placebo (N=14)
Oedema (General disorders) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 764198 20 mg (N=18) | BI 764198 40 mg (N=15) | BI 764198 80 mg (N=15) | Placebo (N=14)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0 | 0
Lenticular opacities (Eye disorders) | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Oral mucosa haematoma (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0
Crying (General disorders) | 0 | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 3 | 0 | 1
Oedema (General disorders) | 1 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 2 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Sense of oppression (General disorders) | 1 | 0 | 0 | 0
Tenderness (General disorders) | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 2
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 2
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Amylase increased (Investigations) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 1 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0
Electrocardiogram ST segment abnormal (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram T wave abnormal (Investigations) | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 2 | 0
Headache (Nervous system disorders) | 3 | 2 | 1 | 2
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1
Oligomenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Capillary fragility (Vascular disorders) | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 2 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2024-01-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT05213624/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-20): https://cdn.clinicaltrials.gov/large-docs/24/NCT05213624/SAP_001.pdf